CLINICAL TRIAL: NCT01077778
Title: Magnetic Resonance Diagnosis of Pulmonary Embolism: Prospective Evaluation in 280 Patients, With Comparison to Multi-slice CT Angiography
Brief Title: Magnetic Resonance Diagnosis of Pulmonary Embolism
Acronym: IRM-EP
Status: Terminated | Type: Observational
Why Stopped: the number of patients will be included is reach
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Aurélie Guimfack, Department Clinical Research of Developpement
Other Study IDs: P051068
Record Dates: First submitted 2010-02-26; First posted 2010-03-01 (Estimated); Last update posted 2016-01-25 (Estimated); Status verified 2007-03

CONDITIONS: Lung Diseases; Pulmonary Embolism
Keywords: Magnetic Resonance Imaging/methods; Magnetic Resonance Angiography; Perfusion Imaging; Pulmonary Embolism/diagnosis
MeSH Terms: conditions — Lung Diseases; Pulmonary Embolism; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Gadolinium-enhanced Magnetic Resonance Imaging — Gadolinium-enhanced Magnetic Resonance Imaging

SUMMARY:
* The purpose of this study is to evaluate the diagnostic accuracy of thoracic magnetic resonance imaging with gadolinium-enhanced, unenhanced and perfusion sequences in patients with clinically suspected acute pulmonary embolism
* Thoracic CT angiography (CTA) will serve as reference standard
* Result of MRI will not interfere with patients' management
* Untreated patients with negative CTA will have 3-month follow-up to verify they were free of thrombose-embolic disease

DETAILED DESCRIPTION:
Background In patients with clinically suspected pulmonary embolism (PE)°with a contraindication to thoracic CT angiography, there is a need for an alternative diagnostic procedure. MRI has not been fully evaluated in this field; moreover, recent technological advances make it necessary to re-evaluate its performance for PE diagnosis.

Design Prospective monocentric study

* Patients with clinically suspected acute pulmonary embolism will undergo thoracic magnetic resonance imaging if inclusion criteria are fulfilled.
* A non-inclusion register will be establish for patients fulfilling the inclusion criteria , not included because MRI was not available (off-hours presentation , another patients already included in the protocol on the same day )

Estimated enrolment : 280 (based on a 25% prevalence of PE in our institution and an expected 80% sensitivity of MRI) Study start date: June 2007 Estimated study completion date: 17 months later (40 to 50 presentations for PE suspicion each month, 20 inclusions expected per month)

Magnetic Resonance imaging: performed on a 1.5 Tesla unit with 3 different sequences

* Unenhanced Steady State Free Precession (SSFP) sequences
* Perfusion imaging following Gadolinium injection at a rate of 5 c/s and a dose of 0.1mmol/kg
* Magnetic resonance angiography following an injection of 0.1mmol/kg of gadolinium at 3ml/s MRI studies will be interpreted secondarily by 2 independent radiologists, blinded to CTA results and clinical probability.

Two different readings will be performed, one global reading and one reading of each sequence separately, displayed in a random order (access base)

Objectives

* to evaluate MRI performance for PE diagnosis globally
* to evaluate the diagnostic value for each sequence (especially the negative predictive value of a normal perfusion sequence)
* to evaluate inter-observer agreement

MRI and CTA have to be performed within 24 hours

ELIGIBILITY:
Inclusion Criteria:

* Clinically suspected acute pulmonary embolism
* 18 years old or more
* D-dimers more than 500 or high clinical probability of pulmonary embolism according to the revised Geneva score
* Thoracic CT angiography performed within 24 hours
* Informed consent

Exclusion Criteria:

* - Contraindication to MRI (pace maker, claustrophobia, any implanted ferromagnetic foreign body)
* Obese patients too large to fit in MRI unit
* Allergy to gadolinium-containing contrast agent or to iodinated contrast media
* Renal insufficiency (clearance less than 30 ml/mn)
* Anticoagulation at a curative dose started more than 48 hours prior to MRI
* Life expectancy less than 3 months
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with acute pulmonary embolism suspicion who fulfil the inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2007-03; Primary Completion 2007-09 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
MRI studies will be interpreted at the end of the inclusion process. CTA results will serve as reference standard to evaluate MRI sensitivity, specificity, positive and negative predictive values. Inter-observer agreement will be evaluated | 17 months after the first inclusion

SECONDARY OUTCOMES:
3 months clinical follow-up will be performed in patients with negative CTA results who did not receive anticoagulation. This is to verify there were no false negatives on CTA | 3 months afer CTA

CONTACTS AND LOCATIONS:
Overall Officials: Marie-pierre Revel, PH, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hopital George Pompidou, Paris, France

REFERENCES:
- [Background] Blum A, Bellou A, Guillemin F, Douek P, Laprevote-Heully MC, Wahl D; GENEPI study group. Performance of magnetic resonance angiography in suspected acute pulmonary embolism. Thromb Haemost. 2005 Mar;93(3):503-11. doi: 10.1160/TH04-08-0495. PMID 15735802
- [Background] Pleszewski B, Chartrand-Lefebvre C, Qanadli SD, Dery R, Perreault P, Oliva VL, Prenovault J, Belblidia A, Soulez G. Gadolinium-enhanced pulmonary magnetic resonance angiography in the diagnosis of acute pulmonary embolism: a prospective study on 48 patients. Clin Imaging. 2006 May-Jun;30(3):166-72. doi: 10.1016/j.clinimag.2005.10.005. PMID 16632150
- [Derived] Revel MP, Sanchez O, Lefort C, Meyer G, Couchon S, Hernigou A, Niarra R, Chatellier G, Frija G. Diagnostic accuracy of unenhanced, contrast-enhanced perfusion and angiographic MRI sequences for pulmonary embolism diagnosis: results of independent sequence readings. Eur Radiol. 2013 Sep;23(9):2374-82. doi: 10.1007/s00330-013-2852-8. Epub 2013 May 8. PMID 23652845